CLINICAL TRIAL: NCT02430649
Title: Irreversible Electroporation(IRE) For Unresectable Prostatic Neoplasms: Phase I and Phase II Clinical Trial
Brief Title: Irreversible Electroporation(IRE) For Unresectable Prostatic Neoplasms
Acronym: IRE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prostatic Neoplasms-IRE-01
Record Dates: First submitted 2015-04-26; First posted 2015-04-30 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Prostatic Neoplasms
Keywords: irreversible electroporation; Unresectable Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IRE Group (Experimental): irreversible electroporation for Unresectable Prostatic Neoplasms
  Interventions: Procedure: Irreversible electroporation (IRE); Device: NanoKnife
- Control (No Intervention): The patients without treatment

INTERVENTIONS:
Procedure: Irreversible electroporation (IRE)
  Other Names: NanoKnife
  Arms: IRE Group
Device: NanoKnife
  Arms: IRE Group

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of irreversible electroporation (IRE) for unresectable Prostatic Neoplasms.

DETAILED DESCRIPTION:
By enrolling patients with unresectable Prostatic Neoplasms adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of percutaneous IRE for unresectable Prostatic Neoplasms.

ELIGIBILITY:
Inclusion Criteria:

* Prostatic Neoplasms diagnosed by positive biopsy or non-invasive criteria,
* Not suitable for surgical resection,
* Eastern Cooperative Oncology Group (ECOG) score of 0-1,
* A prothrombin time ratio > 50%,
* Platelet count > 80x10^9/L,
* Ability of patient to stop anticoagulant and anti-platelet therapy for seven days prior to and seven days post NanoKnife procedure,
* Able to comprehend and willing to sign the written informed consent form (ICF),
* Have a life expectancy of at least 3 months.

Exclusion Criteria:

* Cardiac insufficiency, ongoing coronary artery disease or arrhythmia,
* Any active implanted device (eg Pacemaker),
* Women who are pregnant or women of child-bearing potential who are not using an acceptable method of contraception,
* Have received treatment with an investigational agent/ procedure within 30 days prior to treatment with the NanoKnife™ LEDC System,
* Are in the opinion of the Investigator unable to comply with the visit schedule and protocol evaluations.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-05-20 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse events | 6 month

SECONDARY OUTCOMES:
Percentage of lesions that show no sign of recurrence 12 months after IRE | 12 months
Voltage (A minimum and maximum range of voltage for safe and effective IRE) | 3 months
  A minimum and maximum range of voltage for safe and effective IRE will be analyzed for optimal choice.
Progress free disease (PFS) | 12 months
Overall survival (OS) | 36 months
  Patients will be followed for 36 months after IRE for OS analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Niu, PhD, Study Chair — Fuda Cancer Hospital
Locations (1):
- Biological treatment center in Fuda cancer hospital, Guangzhou, Guangdong, China